CLINICAL TRIAL: NCT02282618
Title: Effects of Cardiac Sympathetic Blockade in Patients With Chronic Heart Failure, a 2-year, Prospective, Randomized Cohort Study
Brief Title: Effects of Cardiac Sympathetic Blockade in Patients With Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Wei Liu, Prof., Harbin Medical University
Other Study IDs: doctorliuwei
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Heart Failure
Keywords: Cardiac Sympathetic Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- heart failure with HTEA: Heart failure patients are treated with the world-wide accepted medicine, plus HTEA for 4 weeks.
- heart failure with medicine: Heart failure patients are treated with the world-wide accepted medicine.
  Interventions: Device: Cardiac Sympathetic Blockade

INTERVENTIONS:
Device: Cardiac Sympathetic Blockade
  Groups: heart failure with medicine

SUMMARY:
Although current pharmaceutical therapies have improved the survival rate in heart failure it remains a fatal disease and is associated with a poor 3-year survival. Increased sympathetic activity found in patients with heart failure plays an important role in the pathogenesis and development of the disease[Provide reference]. Excessive activation of sympathetic tone contributes to arrhythmogenesis, increased cardiac wall tension, and platelet aggregation, promoting a "vicious cycle[What cycle? Elaborate. ]" in these patients.

High thoracic epidural anesthesia (HTEA) can reversibly and regionally block the cardiac sympathetic nervous system. The method was pioneered by Prof. Liu Fengqi in 1995, and he has accumulated clinical experiences from thousands of cases. His anecdotal experience indicates that the method can favorably improve intractable angina, dilated cardiomyopathy, and advanced heart failure. Though the method has been used to treat patients at our center for many years, there has been no prospective trial of its effects on cardiovascular function, or its efficacy to improve clinical outcomes.

The investigators propose to investigate the immediate physiologic effect and clinical effectiveness of HTEA in treating heart failure.

DETAILED DESCRIPTION:
Although current pharmaceutical therapies have improved the survival rate in heart failure it remains a fatal disease and is associated with a poor 3-year survival. Increased sympathetic activity found in patients with heart failure plays an important role in the pathogenesis and development of the disease[Provide reference]. Excessive activation of sympathetic tone contributes to arrhythmogenesis, increased cardiac wall tension, and platelet aggregation, promoting a "vicious cycle[What cycle? Elaborate. ]" in these patients.

High thoracic epidural anesthesia (HTEA) can reversibly and regionally block the cardiac sympathetic nervous system. The method was pioneered by Prof. Liu Fengqi in 1995, and he has accumulated clinical experiences from thousands of cases. His anecdotal experience indicates that the method can favorably improve intractable angina, dilated cardiomyopathy, and advanced heart failure. Though the method has been used to treat patients at our center for many years, there has been no prospective trial of its effects on cardiovascular function, or its efficacy to improve clinical outcomes.

The investigators propose to investigate the immediate physiologic effect and clinical effectiveness of HTEA in treating heart failure.

Methods and design The investigators propose a double-blind placebo-controlled clinical trial. 230 chronic heart failure patients with the course of more than three months will be randomly allocated two groups, 90 in HTEA group, 90 in sham-HTEA (SHAM) group. The investigators will compare their outcomes to 50 historical controls (CON). Ethical approval from our institutional review board will be obtained. Patients will be consented appropriately, and be free to withdraw from the study at any time.

According to the guidelines for chronic heart failure treatment, diuretics, angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, beta-blockers, aldosterone receptor antagonists, digitalis, and vasodilating agents should be used as standard treatments for heart failure in the three groups.

Outcome assessments will be performed objectively by evaluators who have no knowledge of the treatment assignment.

HTEA procedure Patients of HTEA group will be treated with both conventional medical therapy and four weeks of HTEA. The HTEA procedure is as follows: an epidural catheter is inserted through one of the second to fifth thoracic interspaces. Three to five milliliters of 0.5% lidocaine every 2 h are administered to induce a blockade of the cardiac sympathetic segments (Th1-Th5). The catheter remains in place with the lidocaine infusing continuously over the subsequent four weeks.

Sham procedure Patients in the SHAM group will be treated with both conventional medical therapy and four weeks of sham-HTEA. SHAM group received the similiar procedure as HTEA group, except for the infusion of saline water rather than lidocaine..

CON group receive only conventional standard treatment. [For your first trial these outcomes are too ambitious. Just do some initial physiologic experiments first to understand what happens to CHF pts when you perform HTEA. Then follow those pts for the next few weeks]Primary end points[I would first start with short term outcomes. One could use a model such as that outlined in the levosimendan trial http://heartfailure.onlinejacc.org/article.aspx?articleid=1671253 ]: Re-hospitalizing rate caused by severe cardiac failure[Over what time? I would suggest 4 weeks], re-hospitalizing rate caused by other cardiovascular diseases; NYHA cardiac function grading, living quality evaluation, 6 minute walking distance, echocardiography,[When? At 24 hours, at 4 weeks?] dynamic[Is this the same as an ETT?] electrocardiogram, as well as the peripheral blood NT-proBNP [At 24 hrs? 48 hrs? 4 weeks?]changes would be compared. [The statistical plan is missing. Is 50 pts adequate to evaluate the early efficacy.

Potentially see the levosimendan trial to power your study too.

Their methods were as follows:

"The sample size for the REVIVE II trial was estimated on the basis of the following assumptions: the proportion of patients considered improved during the first 5 days would be 50% greater in the levosimendan group than in the placebo group; the proportion of patients considered worse during the first 5 days would be 33% lower in the levosimendan group than in the placebo group; the expected rates of improvement and deterioration in the placebo group would both be 25%; and the study would have >90% power to detect a treatment difference (α = 0.05)."]

Efficacy indicator blood pressure+heart rate+blood oxygen Echocardiography, left ventricular ejection fraction, LVEDd NT-proBNP New York Heart Association functional classification 6-min walking distance quality of life MRI of the heart Safety indicator adverse effect evaluation sheet[Including site-specific problems such as infection]

Baseline 48 hours 1 week 4 weeks 8 weeks Vital signs Echo BNP NYHA class 6 min walk QoL

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure patients with the course of more than three months.

Exclusion Criteria:

* Vavular heart diseases.

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: heart failure
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
mortality | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Harbin Medical University, Harbin, Heilongjiang, China